CLINICAL TRIAL: NCT01379950
Title: The Role of Macrophages in the Inflammatory Resolution Phase in Periodontal Patients
Brief Title: Role of Macrophage in Inflammation Resolution in Periodontal Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Jacob (Cobi) Ekstein - principal investigator, Hadassah Medical Organization
Other Study IDs: perio1-HMO-CTIL
Record Dates: First submitted 2011-05-25; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- periodontitis: patients diagnosed with periodontal disease

SUMMARY:
There is a growing body of evidence to suggest that the resolution of an inflammatory reaction is an active process. This process requiring signals that turn off early inflammatory stages, as neutrophil infiltration and promote resolution phase, as clearance of apoptotic cells. In this array,the relationship between neutrophils, monocytes, and macrophages is crucial for the concert process.

Macrophages possess a plasticity of phenotype that explains their protective as well as potentially detrimental role in chronic inflammation and tissue injury. Such heterogeneity arises as macrophages differentiate from monocytes and are exposed to specific tissue- and hematopoietic cell-derived stimuli. It is important to be able to identify the different types of macrophages in this setting. Today's literature can distinguish between 3 main phenotypic groups of macrophages. The classically activated M1 macrophages, the alternatively activated-M2 macrophages and the "resolution phase" - rMs macrophages. The third phenotypic macrophage might play a crucial rule in the resolution phase, and is called the "resolving macrophage".

All of those pro-resolving lipid mediators promote the return to tissue homeostasis .

The investigators hypothesis is that in periodontal patients the inflammatory process continues because the process does not reach the resolution phase, and in that milieu, the macrophage might be a key component.

Within the overall concept of periodontal disease as a model for an inflammatory disease with an stoppable inflammatory reaction, the primary aim of the study is to check the macrophage characteristics in periodontal patients and to compare it to healthy people.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more, male & female
* generally healthy
* does not take medicine on a regular basis
* has a periodontal disease. control - without a periodontal disease
* no periodontal treatment for at list 6 months prior to his acceptance to the trail
* willing to donate 50 ml of blood twice during the trail
* understands the trail and gave a consent to participate

Exclusion Criteria:

* pregnancy or nursing
* chronic use of alcohol
* systemic conditions - diseases, neoplastic lesions in the oral cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients coming to the periodontal clinic in the dental school in order to attend a periodontal treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
The macrophage phenotype (M1, M2, resolution phase macrophage) | 1 year
  we will try to specify the characteristics of the macrophage phenotype and to see whether there is a difference between periodontal patients and healthy ones.

CONTACTS AND LOCATIONS:
Locations (1):
- Periodontal Clinic, Faculty of Dental Medicine, Hebrew University and Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Bystrom J, Evans I, Newson J, Stables M, Toor I, van Rooijen N, Crawford M, Colville-Nash P, Farrow S, Gilroy DW. Resolution-phase macrophages possess a unique inflammatory phenotype that is controlled by cAMP. Blood. 2008 Nov 15;112(10):4117-27. doi: 10.1182/blood-2007-12-129767. Epub 2008 Sep 8. PMID 18779392